CLINICAL TRIAL: NCT05037214
Title: Measure of Stress After the First Wave of Covid 19 Within Hospital Workers
Brief Title: COVID-19 : Stress Within Hospital Workers
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0548
Record Dates: First submitted 2021-09-06; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: COVID 19; Depression; Stress, Psychological; Burnout
Keywords: Psychiatry; Healthcare staff
MeSH Terms: conditions — COVID-19; Depression; Stress, Psychological; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As of December 2019, the global pandemic of COVID-19 has spread rapidly throughout the world, putting healthcare staff at the frontline.

In this context, several factors leading to the appearance of psychiatric symptoms have emerged : work overload, fear of being infected or of infecting, exhaustion… (The Lancet, 2020)

Indeed, post-traumatic stress disorder (PTSD), depressive symptoms, anxiety symptoms, insomnia and increased stress have been reported (Rossi et al., 2020).

Furthermore, the increased anxiety and depression symptoms and stress associated with the COVID-19 pandemic may increase the risk of suicide in this already high-risk population. For example, suicidal ideation has been reported in up to 5% of healthcare workers in the United States (Young et al., 2021).

It is therefore essential to evaluate the incidence of psychiatric disorders (e.g. PTSD, depression, suicide) and their associated risk factors among the hospital staff.

To do so, Montpellier University Hospital healthcare staff was asked their mental state during the first wave of COVID-19.

ELIGIBILITY:
Inclusion criteria:

* Healthcare staff working at Montpellier University Hospital during the first wave of COVID-19
* Having responded to the online survey sent to all healthcare staff

Exclusion criteria:

- Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare staff working during the first wave of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 779 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms | day 1
  anxiety level assessed with the Generalized Anxiety Disorder questionnaire (GAD-7) : higher score indicates higher anxiety (min : 0; max : 21)
Depression symptoms | day 1
  depression symptomatoloy assessed with the Patient Health Questionnaire (PHQ-9) : higher score indicates higher depression level (min : 0; max : 27)
Sleep | day 1
  sleep quality assessed with the Insomnia Severity Index (ISI) : higher score indicates higher insomnia level (min : 0; max : 28)

SECONDARY OUTCOMES:
Post traumatic stress disorder | day 1
  post traumatic stress disorder symptomatology assessed with the Posttraumatic stress disorder Checklist Scale (PCL-S) : higher score indicates more sever post traumatic stress disorder symptoms
Physical pain | day 1
  physical pain assessed with a likert scale
Burnout symptoms | day 1
  burnout symptomatology assessed with the Maslach Burnout Inventory (MBI) : higher scores on the emotional exhaustion scale and the depersonalization scale and lower score on the professional accomplishment scale indicate higher burnout level.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte NOBILE, PharmD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC